CLINICAL TRIAL: NCT04298372
Title: Frontline Lenalidomide for AL Amyloidosis Involving Myocardium: Investigation of Organ Reversing Capacity of Lenalidomide
Brief Title: Frontline Lenalidomide for AL Amyloidosis Involving Myocardium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, YOUNGIL KOH, Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1810-089-981
Record Dates: First submitted 2019-12-03; First posted 2020-03-06 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Amyloidosis Cardiac
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Lenalidomide 25mg — As single arm study, patients will be treated as follows:
  * Lenalidomide : D1~D21 daily oral administration, starting dose 15mg, with an increase of 5mg every cycle, if tolerated, up to 25mg.
  * Dexamethasone : D1~D4 daily oral administration or intravenous injection, 40mg(or 20mg for age for age ≥ 65 years old) Patients will be treated every 4 weeks as one cycle, and up to 12 cycles of treatment will be conducted.
  Other Names: Revlimid 25mg

SUMMARY:
This phase II clinical trial aimed at influencing the improvement of major organ functions, especially the objective response rate, in Amyloid light-chain amyloidosis involving myocardium.

DETAILED DESCRIPTION:
This study was designed according to the 18F-florbetaben positron emission tomography imaging, which successfully demonstrated a significant reduction in the amount of amyloid in the heart when administered by merging thalidomide and dexamethasone in patients involving myocardium, and reported that this reaction leads to an improvement in cardiac function. Amyloid light-chain amyloidosis patients at age 19 or older with refractory or relapsed who participants should have never been exposed to lenalidomide within 5 years. Planned initial dosage of the current regimen are as follow;

* Lenalidomide : D1~D21 daily oral administration, starting dose 15mg, with an increase of 5mg every cycle, if tolerated, up to 25mg.
* Dexamethasone : D1~D4 daily oral administration or intravenous injection, 40mg(or 20mg for age for age ≥ 65 years old) Patients will be treated every 4 weeks as one cycle, and up to 12 cycles of treatment will be conducted. The investigator is working on a total of 30 patients, the primary endpoint of this study is objective response rate and secondary endpoints are cardiac/renal/hepatic function, 18F-florbetaben positron emission tomography imaging parameter, overall survival period, progression-free survival period, toxicity profile.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 19 years old
* Amyloid light-chain amyloidosis patients who meet both(A and B) of the following criteria

A. Cardiac involvement: meet one or more of the following criteria

1. Echocardiography : mean wall thickness > 12mm, and no other cardiac cause
2. Cardiac MRI : CMR was considered positive for amyloid cardiomyopathy if there were morphologic and structural abnormalities consistent with the diagnosis (wall thickening of the left ventricular [LV], right ventricular [RV], or interatrial septum and biatrial enlargement) coupled with abnormal myocardial nulling and diffuse or irregular delayed gadolinium enhancement of the LV myocardium.
3. N-terminal prohormone of brain natriuretic peptide : > 332ng/l in the absence pf renal failure

B. Exposure history to lenalidomide: participants should have never been exposed to lenalidomide within 5 years.

* Eastern Cooperative Oncology Group performance status ≤ 3
* Patients must meet the following clinical laboratory criteria with 2 weeks of starting treatment:

  1. Serum creatinine ≤ 3.0mg/dl or Creatinine Clearance ≥ 50ml/minute (Cockcroft-Gault)
  2. Absolute neutrophil count ≥ 1000/ul
  3. Platelet ≥ 75,000/ul
  4. Hemoglobin ≥ 8.0mg/dl
  5. Bilirubin < 2 times or Alkaline phosphate < 4 times upper limit of normal
* At least 3 months of existence are expected from the time of enroll this study
* A female of childbearing potential(is defined as a sexually mature woman who: 1 has not undergone a hysterectomy or bilateral oophorectomy or 2, has not been naturally post-menopausal (amenorrhea following cancer therapy does not rule out childbearing potential) must have a negative pregnancy test prior to treatment.

  1. must agree to use two reliable methods of contraception simultaneously or practice complete abstinence from any heterosexual intercourse during the following time periods related to this study: for at least 4 weeks after study treatment discontinuation.
  2. must have two(serum and urine) negative pregnancy test during screening period
  3. must have serum and urine negative pregnancy test within 10-14 days and 24hrs before commencing lenalidomide
* Male patients who agree to practice effective barrier contraception during the entire study treatment period and through 30 days after the last dose of study treatment
* Patients who understand and voluntarily agree to the contents of the research statement in writing and who are willing and able to comply with the visit schedule, treatment plan, laboratory examination and other testing procedures

Exclusion Criteria:

* Amyloid light-chain amyloidosis without cardiac involvement
* Patients who are planning to receive autologous stem cell transplantation or received autologous stem cell transplantation, remained in hematologic complete response
* Pregnant, lactating or unwilling to use adequate contraception
* Male patients who unwilling to practice effective barrier contraception during the entire study treatment period and through 30 days after the last dose of study treatment
* Patients with acute infections requiring nonpermanent therapy (antibiotics, antibacterial drugs, or antiviral drugs) within 14 days of the first administration of the lenalidomide or with a history of systemic fungal infections and infections without valid antimicrobial agents
* Any clinically significant history of genetic, kidney, neurological, psychiatric, endocrine, metabolism, immunological, cardiovascular, lung, or liver diseases in the investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent.
* Patients with known history of allergic and hypersensitivity for investigational product, their analogous bodies, or the subtypes contained in the various forms of any preparation
* Patients who were given a live vaccine within 8 weeks of the first dose of the drug
* Chemotherapy with approved or investigation anticancer therapeutics within 4 weeks prior to starting this study
* Patients who are unable to voluntarily agree to participate in a study or who are not willing to participate

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | After completion of 12 cycles of treatment(each cycle is 28 days)
  ORR is defined as the percentage of subjects with evidence of a confirmed CR(complete response), VGPR(very good partial response) or PR(partial response)

SECONDARY OUTCOMES:
Change of the cardiac function | At Baseline and the end of each 1-12 cycles (baseline and 1-12 months)
  Change of the cardiac function will be observed with the NTproBNP levels.
Change of the renal function | At Baseline and the end of each 1-12 cycles (baseline and 1-12 months)
  Change of the renal function will be observed with the 24h urine protein levels.
Change of the hepatic function | At Baseline and the end of each 1-12 cycles (baseline and 1-12 months)
  Change of the hepatic function will be observed with the alkaline phophatase levels.

CONTACTS AND LOCATIONS:
Overall Officials: Youngil Koh, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No